CLINICAL TRIAL: NCT01623830
Title: Targeting Memory Reconsolidation to Prevent the Return of Fear in a Pilot Randomized Clinical Trial
Brief Title: Targeting Reconsolidation to Prevent Return of Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Barbara O. Rothbaum, PhD, Professor in Psychiatry and Associate Vice Chair of Clinical Research, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00056442; Reconsolidation_NIMH_2012 (Other: Other)
Record Dates: First submitted 2012-06-12; First posted 2012-06-20 (Estimated); Results first posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Fear of Flying
Keywords: reconsolidation; fear of flying; virtual reality; virtual reality exposure therapy
MeSH Terms: conditions — Aerophobia | interventions — Virtual Reality Exposure Therapy; Implosive Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reactivation + VRE (Experimental): Virtual reality exposure therapy (VRE) for the fear of flying (FOF) preceded by a reminder of the feared stimulus (a virtual reality clip of a virtual airplane taxiing and taking off) presented in the head mounted display 10 minutes prior to all VR exposure therapy sessions
  Interventions: Behavioral: Virtual Reality Exposure Therapy
- Neutral Cue + VRE (Active Comparator): VRE for the FOF preceded by a neutral cue (a virtual reality clip of a virtual living room) presented in the head mounted display 10 minutes prior to all VR exposure therapy sessions.
  Interventions: Behavioral: Virtual Reality Exposure Therapy

INTERVENTIONS:
Behavioral: Virtual Reality Exposure Therapy — Treatment will consist of 8 weekly sessions. Session 1: information gathering, treatment procedures and rationale. Session 2: Cognitive restructuring. Session 3: Breathing retraining and thought stopping. Session 4: Review cognitive restructuring and hyperventilation exposure. Sessions 5-8 Fear of flying exposure in the Virtual environment.
  Other Names: exposure therapy; fear of flying treatment

SUMMARY:
The overall aim of this project is to determine if using a cue to trigger (and reactivate) the fear memory 10 minutes prior to exposure treatment sessions leads to less anxiety in patients with a fear of flying. The long term goals are to establish if targeting the reconsolidation of fear with a reminder of the fear is effective for human clinical populations in reducing relapse (return of fear). In this investigation, the investigators propose to treat 64 patients diagnosed with a fear of flying (FOF) using virtual reality exposure therapy (VRE). All patients in the study will receive exactly the same exposure treatment using a virtual airplane.

DETAILED DESCRIPTION:
Prior to each VRE session, the investigators will test a brief, easy-to-implement manipulation that triggers the fear memory and presumably allows it to be changed in a way that prevents the fear from returning later (i.e., prevents relapse). The investigators propose to randomly assign eligible participants to 1 of 2 conditions: 1) VRE therapy preceded by a reminder of the feared stimulus (a VR clip of a virtual airplane taxiing and taking off) presented 10 minutes prior to all VRE therapy sessions, or 2) VRE therapy preceded by a neutral cue (a VR clip of a virtual living room) presented 10 minutes prior to all VRE therapy sessions. Participants will be evaluated pre- and post-treatment and at a 3 month and 6 month follow-up visit to assess long-term effects.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants, male and female, ages 18-70;
2. Participants must meet Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria for specific phobia, situational type or panic disorder with agoraphobia, in which flying is the primary feared stimulus, or agoraphobia without a history of panic disorder, in which flying is a feared stimulus; Participants may have comorbid depression or anxiety disorders to increase generalizability of sample, but fear of flying must be the primary complaint;
3. Participants must have flown at least once before;
4. Participants on psychoactive medications must be stabilized on that dose and medication for at least three months, and must agree to remain on that dose throughout the project. All assessments will include a form inquiring about any medication changes, and participants on medications will be monitored by their prescribing physician; and
5. Participants must be literate in English.

Exclusion Criteria:

1. Patients with current or history of mania, schizophrenia, or other psychoses;
2. Patients with current (past 3 months) prominent suicidal ideation;
3. Patients with current alcohol or drug abuse/dependence; and
4. Patients unable to wear the virtual reality head mounted display for any reason (i.e. due to panic disorder, head discomfort, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2012-07; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara O Rothbaum, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reactivation + VRE | Neutral Cue + VRE
Started | 45 | 44
Completed | 38 | 35
Not Completed | 7 | 9
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Exclusion from Study | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reactivation + VRE | Neutral Cue + VRE | Total
Number analyzed (Participants) | 45 | 44 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 44 | 89
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 37 | 34 | 71
  Male | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 45 | 44 | 89

OUTCOME MEASURES:

1. Primary Outcome: Fear of Flying Inventory (FFI)
Description: a 33-item scale measuring intensity of FOF. Items are rated on a 9-point scale ranging from 0 ( not at all) to 8 ( very severely disturbing). The possible range of scores is 0-264 with higher total scores indicating greater fear of flying intensity.Test-retest reliability for 15 WL patients was .92, and it has been sensitive to change with treatment.
Time Frame: Post treatment (9 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reactivation + VRE | Neutral Cue + VRE
Number analyzed (Participants) | 38 | 35
units on a scale | 65.55 (49.88) | 76.57 (47.46)

2. Primary Outcome: The Questionnaire on Attitudes Toward Flying (QAF)
Description: assesses history of FOF, previous treatment, and attitudes toward flying. It includes a 36-item questionnaire rating the level of fear on an 11-point scale ranging from 0 to10 in different flying situations. The possible range of scores is 0 to 360 with higher scores indicating greater fear associated with flying. Test-retest reliability was .92, and split-half reliability was .99.
Time Frame: post treatment (9 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reactivation + VRE | Neutral Cue + VRE
Number analyzed (Participants) | 38 | 35
units on a scale | 126.29 (85.32) | 123.46 (66.87)

3. Secondary Outcome: The Beck Depression Inventory (BDI)
Description: a 21-item measure of cognitive and vegetative symptoms of depression is widely used in a variety of populations, including trauma victims and is sensitive to treatment effects on depression. The possible range for scores is 0-63 with higher scores suggesting more severe symptoms of depression.
Time Frame: post-treatment (9 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reactivation + VRE | Neutral Cue + VRE
Number analyzed (Participants) | 38 | 35
units on a scale | 4.26 (5.39) | 3.6 (3.74)

4. Secondary Outcome: State Trait Anxiety Inventory- State (STAI-State)
Description: The STAI-State is a 20-item self report scale employing a Likert scale format with 4 responses per item (1-4). The possible range of scores is from 20-80, and higher scores indicate greater levels of anxiety.Ten of the STAI items measure feelings of stress and anxiety, while the remaining ten items measure feelings of relaxation.
Time Frame: post-treatment (9 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reactivation + VRE | Neutral Cue + VRE
Number analyzed (Participants) | 38 | 35
units on a scale | 45.97 (5.05) | 46.29 (5.40)

5. Secondary Outcome: State Trait Anxiety Inventory- Trait (STAI-Trait)
Description: The STAI-Trait is a 20-item self report scale employing a Likert scale format with 4 responses per item (1-4). The possible range of scores is from 20-80, and higher scores indicate greater levels of anxiety. Ten of the STAI items measure feelings of stress and anxiety, while the remaining ten items measure feelings of relaxation.
Time Frame: post-treatment (9 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reactivation + VRE | Neutral Cue + VRE
Number analyzed (Participants) | 38 | 35
units on a scale | 44.83 (4.36) | 45.81 (4.18)

ADVERSE EVENTS:
Arm/Group | Reactivation + VRE | Neutral Cue + VRE
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 0/45 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes